CLINICAL TRIAL: NCT06815081
Title: A Study to Determine a Capillary Alternative to the Gold Standard Oral Glucose Tolerance Test
Brief Title: Capillary OGTT Study
Acronym: CapOGTT
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: University of Bristol (Other); Yale University (Other); Oxford University Hospitals NHS Trust (Other); Nottingham University Hospitals NHS Trust (Other); Cardiff and Vale University Health Board (Other Government); Royal London Hospital, Barts Health NHS Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: PID16905
Record Dates: First submitted 2025-01-27; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: Capillary; Glucose; Oral glucose tolerance test; Method Comparison; Feasibility; Acceptability; Type 1 diabetes; Monitoring; Follow-up; Screening
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1 (Simultaneous venous and capillary OGTT): To assess the ability of the capillary OGTT to be a reliable and acceptable alternative to the standard venous OGTT in children, investigators will aim to capture a spread of glucose values across the whole diagnostic range.
  This will be undertaken in clinical and research settings, led by either a healthcare professional or research nurse.
  Children undergoing a standard venous OGTT will be invited to complete a capillary OGTT. Both venous and capillary samples will be collected at the same time. Investigators will also invite children with stage 3 (clinical) T1D to capture glucose levels in the hyperglycaemic range. These participants will receive a smaller glucose dose for their OGTT (1g/kg, max dose 75g), to attenuate their glucose rise and allow the comparison of clinically meaningful glucose values. Participants will be asked to complete a questionnaire following the OGTT to obtain information about acceptability.
- Cohort 2 (Capillary OGTT at home): In this cohort (running concurrently alongside cohort 1) investigators aim to assess the acceptability and feasibility of a capillary OGTT device in children and young people with early-stage (known stage 1 or 2) T1D.
  This will take place in the home of participants, with written and video instructions provided.
  Children known to be positive for ≥ 2 IAb will be invited to take part and will be sent a capillary OGTT test kit which will include a glucose drink, lancets and instructions (written and video).
  They will fast overnight (from midnight the night before, for a minimum of 8 hours) before completing a 2-hour OGTT using the test kit and instructions provided. Glucose samples will be collected at 0 and 120 minutes. Participants will be asked to complete a questionnaire following completion of the OGTT, to obtain information about acceptability.
- Cohort 1 (CGM sub-study): In this sub-study investigators aim to explore the ability of CGM to be an alternative to the standard venous OGTT. A subgroup of participants in cohort 1 with known T1D (stage 1, 2 or 3) will be invited to wear a CGM sensor for up to 10 days, which will be worn during their OGTT, at home during a standard mixed meal and free-living.
  Whilst wearing the CGM at home, participants will be asked to consume a liquid mixed meal (Ensure Plus, 6ml/kg maximum 360ml, preceded by an 8-hour fast) and complete a 3-day food diary, by photographing the largest meal of the day to allow estimation of carbohydrate intake (not the same day as the OGTT or liquid mixed meal). Participants will then be asked to complete a questionnaire to obtain information about acceptability.
- Qualitative sub-study: To understand the factors that contribute to uptake of monitoring offered to children at risk of type 1 diabetes, investigators will invite a small number of young people (aged 15-18) and parents to take part in a semi-structured interview. Investigators will also invite healthcare professionals involved in delivering metabolic testing as part of follow-up to take part in semi-structured interviews, to understand their views on the factors which may influence future implementation into clinical care.

SUMMARY:
Type 1 diabetes (T1D) is a chronic condition, affecting 1 in 490 children under the age of 15 years. It is caused by the immune system damaging the pancreas, the organ which makes insulin. T1D has recognised stages before symptoms develop, providing an opportunity for early diagnosis, education and treatment which may delay the onset of symptoms. Early diagnosis often relies on a test called the oral glucose tolerance test (OGTT), which is commonly used but not well tolerated, possibly because it requires a drip inserted into the vein, and several blood samples taken over 2-3 hours in a healthcare setting.

This study aims to test whether an OGTT using a finger-prick to test glucose, can be done at home. This is the 'GTT@home'. The finger-prick creates a drop of blood, which is done before and two hours after drinking a sugary drink. Investigators will also explore whether a continuous glucose monitor (CGM), which reads glucose levels through the skin could be an alternative. The investigators plan to recruit 90 children and young people, across two groups to assess the GTT@home.

To understand the experiences of those involved in monitoring, the investigators will invite young people, parents and healthcare workers to take part in an interview, to understand the impact of testing to predict clinical T1D.

Group 1 will assess the accuracy of measuring glucose from a finger-prick blood test when compared to a blood test from the vein. The investigators will recruit individuals who are having an OGTT as part of a research study, for clinical care, or if individuals have agreed to have an OGTT for this study. Those with T1D will be invited to wear a CGM to explore its use as an additional, practical alternative.

Group 2 will assess how well the GTT@home test works when done at home and how acceptable it is. This will only be offered to those known to be at risk of T1D.

These studies will help investigators to understand if the GTT@home can be used in routine care.

ELIGIBILITY:
Inclusion criteria:

Cohort 1

* Willing and able to give informed consent for participation, or assent with parental consent
* Aged < 18 years old
* Able to consume oral glucose drink within 10 minutes
* Undergoing an OGTT, or consent to have one

Cohort 2

* Positive for two or more islet autoantibodies at any time
* Willing and able to give informed consent for participation, or assent with parental consent
* Aged < 18 years old
* Able to consume oral glucose drink within 10 minutes

CGM sub-study

* Willing and able to give informed consent for participation, or assent with parental consent
* Aged < 18 years old
* Able to consume oral glucose drink within 10 minutes
* Confirmed to have stage 1, 2 or 3 T1D
* Participation in Cohort 1

Qualitative sub-study

* Willing and able to give informed consent for participation, or assent with parental consent Then EITHER
* A young person positive for two or more islet autoantibodies (15 years old and above) at any time, or parent of a young person who has experienced a metabolic test e.g. OGTT OR
* A healthcare professional involved in delivering metabolic testing

Exclusion Criteria:

Cohort 1

* Any known haemoglobinopathy
* Cystic fibrosis related diabetes
* Non-English speaker

Cohort 2

* Any known haemoglobinopathy
* Known clinical diabetes and on treatment
* Non-English speaker
* No recent weight available (within 3 months of study visit) and unable to obtain new weight measurement

CGM sub-study

* Any known haemoglobinopathy
* Cystic fibrosis related diabetes
* Non-English speaker
* Any active skin issue which would prevent the use of a CGM device

Qualitative sub-study

• Non-English speaker

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Cohort 1 - Children < 18 years of age, across a range of ages, will be invited to take part. To get a spread of glucose values, we will aim to recruit approximately equal numbers of participants with normoglycaemia, dysglycaemia and hyperglycaemia.
  Cohort 1 CGM sub-study - Children < 18 years of age, who have T1D stage 1, 2 or 3 and undergoing an OGTT in cohort 1 will be invited to take part.This sub-study will be additional and optional to cohort 1.
  Cohort 2 - Children < 18 years of age, who are identified as having stage 1, 2 or 3 T1D will be invited to take part in an OGTT at home.
  Qualitative sub-study - Young people ≥ 15 years old with T1D stage 1, 2 or recent stage 3 (up to 12 months), who have been involved in metabolic follow-up, will be invited to take part. Parents of a child (of any age) with T1D stage 1, 2 or recent stage 3 will also be invited. Healthcare professionals involved in delivering metabolic follow-up for children with diabetes antibodies will also be invited.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
To determine the agreement of capillary blood glucose levels to venous blood glucose levels during a standard OGTT | From enrolment to end of study visit on day 1.
  Agreement between capillary and blood glucose measures.
To assess the feasibility of using the capillary OGTT device in the home environment | From enrolment to end of study visit on day 1
  1. Proportion of successful glucose readings at 0, 120 minutes
  2. Proportion of errors/missing glucose readings
  3. Proportion of adverse events

SECONDARY OUTCOMES:
To determine the diagnostic accuracy of capillary blood glucose levels at diagnostic thresholds | From enrolment to end of study visit on day 1.
  Sensitivity and specificity of capillary glucose at 5.6mmol/L, 7.0mmol/L (fasting), 11.1 mmol/L (60 min), and 7.8mmol/L and 11.1mmol/L (120 min).
Assess the acceptability of the capillary OGTT device | From enrolment to end of study visit on day 1.
  Acceptability by questionnaire (Parent +/- child), using either a standard 7-point Likert scale (1 - not painful at all, 7 - very painful) for participants aged 16 and above, or Wong Baker Faces pain scale (0 - no hurt, 10 - hurts worst) for participants aged under 16.
To assess the in-depth experience of participants attending study visits involving a metabolic test or assessment | From enrolment to end of study visit on day 1
  Analysis of qualitative interviews from young people.
To assess the in-depth experience of parents attending study visits with their child involving a metabolic test or assessment | From enrolment to end of study visit on day 1.
  Analysis of qualitative interviews from parents.
To assess the in-depth views of healthcare professionals involved in the delivery of a metabolic test or assessment of a child | From enrolment to end of study visit on day 1.
  Analysis of qualitative interviews from healthcare professionals.

OTHER OUTCOMES:
To explore the diagnostic accuracy of CGM to define T1D stages during a standard OGTT | From enrolment to end of study visit at day 10.
  Sensitivity/specificity of sensor glucose levels at diagnostic thresholds.
To explore CGM values at fasting and 120-minutes and its relation to OGTT measures of glucose, during a) standard liquid mixed meal, and b) free-living | From enrolment to end of study visit on day 10.
  Sensor glucose variability (coefficient of variation (%CV)), during home meals, across different T1D stages.
To explore CGM values at fasting and 120-minutes and its relation to OGTT measures of glucose, during a) standard liquid mixed meal, and b) free-living | From enrolment to end of study visit on day 10.
  Sensor glucose variability (mean amplitude of glycaemic excursion (MAGE) mmol/L)), during home meals, across different T1D stages.
To explore CGM values at fasting and 120-minutes and its relation to OGTT measures of glucose, during a) standard liquid mixed meal, and b) free-living | From enrolment to end of study visit on day 10.
  Sensor glucose variability (low blood glucose index (LBGI)), during home meals, across different T1D stages.
To explore CGM values at fasting and 120-minutes and its relation to OGTT measures of glucose, during a) standard liquid mixed meal, and b) free-living | From enrolment to end of study visit on day 10.
  Sensor glucose variability (high blood glucose index (HBGI)), during home meals, across different T1D stages.
To explore CGM values at fasting and 120-minutes and its relation to OGTT measures of glucose, during a) standard liquid mixed meal, and b) free-living | From enrolment to end of study visit on day 10.
  Sensor glucose variability (average daily risk range (ADRR)), during home meals, across different T1D stages.

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Noah's Ark Childrens Hospital for Wales, Cardiff
  - Royal London Barts Health NHS Trust, London
  - Nottingham Childrens Hospital, Nottingham
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Dates of birth will not be shared, but ages (possibly grouped) will be provided.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting information will be availabile once the primary paper for the study has been published.
Access Criteria: Subject to participant consent, data will be shared with other researchers for research projects that have appropriate ethical approval. Requests for access to the data will be controlled by the Data Access Committee.

REFERENCES:
- [Background] Wilson DM, Pietropaolo SL, Acevedo-Calado M, Huang S, Anyaiwe D, Scheinker D, Steck AK, Vasudevan MM, McKay SV, Sherr JL, Herold KC, Dunne JL, Greenbaum CJ, Lord SM, Haller MJ, Schatz DA, Atkinson MA, Nelson PW, Pietropaolo M; Type 1 Diabetes TrialNet Study Group. CGM Metrics Identify Dysglycemic States in Participants From the TrialNet Pathway to Prevention Study. Diabetes Care. 2023 Mar 1;46(3):526-534. doi: 10.2337/dc22-1297. PMID 36730530
- [Background] Ylescupidez A, Speake C, Pietropaolo SL, Wilson DM, Steck AK, Sherr JL, Gaglia JL, Bender C, Lord S, Greenbaum CJ. OGTT Metrics Surpass Continuous Glucose Monitoring Data for T1D Prediction in Multiple-Autoantibody-Positive Individuals. J Clin Endocrinol Metab. 2023 Dec 21;109(1):57-67. doi: 10.1210/clinem/dgad472. PMID 37572381
- [Background] Liu Y, Rafkin LE, Matheson D, Henderson C, Boulware D, Besser REJ, Ferrara C, Yu L, Steck AK, Bingley PJ; Type 1 Diabetes TrialNet Study Group. Use of self-collected capillary blood samples for islet autoantibody screening in relatives: a feasibility and acceptability study. Diabet Med. 2017 Jul;34(7):934-937. doi: 10.1111/dme.13338. Epub 2017 Mar 8. PMID 28226181
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. J Clin Epidemiol. 2008 Apr;61(4):344-9. doi: 10.1016/j.jclinepi.2007.11.008. PMID 18313558
- [Background] Dunseath GJ, Bright D, Luzio SD. Comparative Accuracy Evaluation of a Blood Glucose Meter With Novel Hematocrit Correction Technology, With Three Currently Used Commercially Available Blood Glucose Monitoring Systems. J Diabetes Sci Technol. 2019 May;13(3):568-574. doi: 10.1177/1932296818821389. Epub 2019 Jan 9. PMID 30623673
- [Background] Ginsberg BH. Factors affecting blood glucose monitoring: sources of errors in measurement. J Diabetes Sci Technol. 2009 Jul 1;3(4):903-13. doi: 10.1177/193229680900300438. PMID 20144340
- [Background] Bethel MA, Price HC, Sourij H, White S, Coleman RL, Ring A, Kennedy IE, Tucker L, Holman RR. Evaluation of a self-administered oral glucose tolerance test. Diabetes Care. 2013 Jun;36(6):1483-8. doi: 10.2337/dc12-0643. Epub 2013 Jan 15. PMID 23321216
- [Background] Dunseath GJ, Bright D, Jones C, Dowrick S, Cheung WY, Luzio SD. Performance evaluation of a self-administered home oral glucose tolerance test kit in a controlled clinical research setting. Diabet Med. 2019 Jul;36(7):862-867. doi: 10.1111/dme.13961. Epub 2019 Apr 26. PMID 30972793
- [Background] Bruns DE, Metzger BE, Sacks DB. Diagnosis of Gestational Diabetes Mellitus Will Be Flawed until We Can Measure Glucose. Clin Chem. 2020 Feb 1;66(2):265-267. doi: 10.1093/clinchem/hvz027. No abstract available. PMID 32040567
- [Background] Plebani M. The detection and prevention of errors in laboratory medicine. Ann Clin Biochem. 2010 Mar;47(Pt 2):101-10. doi: 10.1258/acb.2009.009222. Epub 2009 Dec 1. PMID 19952034
- [Background] Bogdanet D, O'Shea P, Lyons C, Shafat A, Dunne F. The Oral Glucose Tolerance Test-Is It Time for a Change?-A Literature Review with an Emphasis on Pregnancy. J Clin Med. 2020 Oct 27;9(11):3451. doi: 10.3390/jcm9113451. PMID 33121014
- [Background] Sosenko JM, Skyler JS, DiMeglio LA, Beam CA, Krischer JP, Greenbaum CJ, Boulware D, Rafkin LE, Matheson D, Herold KC, Mahon J, Palmer JP; Type 1 Diabetes TrialNet Study Group; Diabetes Prevention Trial-Type 1 Study Group. A new approach for diagnosing type 1 diabetes in autoantibody-positive individuals based on prediction and natural history. Diabetes Care. 2015 Feb;38(2):271-6. doi: 10.2337/dc14-1813. Epub 2014 Dec 17. PMID 25519451
- [Background] Simmons KM, Sosenko JM, Warnock M, Geyer S, Ismail HM, Elding Larsson H, Steck AK. One-Hour Oral Glucose Tolerance Tests for the Prediction and Diagnostic Surveillance of Type 1 Diabetes. J Clin Endocrinol Metab. 2020 Nov 1;105(11):e4094-101. doi: 10.1210/clinem/dgaa592. PMID 32844178
- [Background] Sosenko JM, Skyler JS, Palmer JP; Diabetes Type 1 TrialNet and Diabetes Prevention Trial-Type 1 Study Groups. The development, validation, and utility of the Diabetes Prevention Trial-Type 1 Risk Score (DPTRS). Curr Diab Rep. 2015 Aug;15(8):49. doi: 10.1007/s11892-015-0626-1. PMID 26077017
- [Background] Sosenko JM, Skyler JS, Mahon J, Krischer JP, Greenbaum CJ, Rafkin LE, Beam CA, Boulware DC, Matheson D, Cuthbertson D, Herold KC, Eisenbarth G, Palmer JP; Type 1 Diabetes TrialNet and Diabetes Prevention Trial-Type 1 Study Groups. Use of the Diabetes Prevention Trial-Type 1 Risk Score (DPTRS) for improving the accuracy of the risk classification of type 1 diabetes. Diabetes Care. 2014 Apr;37(4):979-84. doi: 10.2337/dc13-2359. Epub 2014 Feb 18. PMID 24550217
- [Background] Bediaga NG, Li-Wai-Suen CSN, Haller MJ, Gitelman SE, Evans-Molina C, Gottlieb PA, Hippich M, Ziegler AG, Lernmark A, DiMeglio LA, Wherrett DK, Colman PG, Harrison LC, Wentworth JM. Simplifying prediction of disease progression in pre-symptomatic type 1 diabetes using a single blood sample. Diabetologia. 2021 Nov;64(11):2432-2444. doi: 10.1007/s00125-021-05523-2. Epub 2021 Aug 2. PMID 34338806
- [Background] Weiss A, Zapardiel-Gonzalo J, Voss F, Jolink M, Stock J, Haupt F, Kick K, Welzhofer T, Heublein A, Winkler C, Achenbach P, Ziegler AG, Bonifacio E; Fr1da-study group. Progression likelihood score identifies substages of presymptomatic type 1 diabetes in childhood public health screening. Diabetologia. 2022 Dec;65(12):2121-2131. doi: 10.1007/s00125-022-05780-9. Epub 2022 Aug 27. PMID 36028774
- [Background] Driscoll KA, Tamura R, Johnson SB, Gesualdo P, Clasen J, Smith L, Jacobsen L, Elding Larsson H, Haller MJ; TEDDY Study Group. Adherence to oral glucose tolerance testing in children in stage 1 of type 1 diabetes: The TEDDY study. Pediatr Diabetes. 2021 Mar;22(2):360-368. doi: 10.1111/pedi.13149. Epub 2021 Jan 6. PMID 33179853
- [Background] Sims EK, Geyer S, Johnson SB, Libman I, Jacobsen LM, Boulware D, Rafkin LE, Matheson D, Atkinson MA, Rodriguez H, Spall M, Elding Larsson H, Wherrett DK, Greenbaum CJ, Krischer J, DiMeglio LA; Type 1 Diabetes TrialNet Study Group. Who Is Enrolling? The Path to Monitoring in Type 1 Diabetes TrialNet's Pathway to Prevention. Diabetes Care. 2019 Dec;42(12):2228-2236. doi: 10.2337/dc19-0593. Epub 2019 Sep 26. PMID 31558546
- [Background] Quinn LM, Swaby R, Tatovic D, Narendran P, Besser REJ, Dayan CM. What does the licensing of teplizumab mean for diabetes care? Diabetes Obes Metab. 2023 Aug;25(8):2051-2057. doi: 10.1111/dom.15071. Epub 2023 Apr 24. No abstract available. PMID 36999237
- [Background] Herold KC, Bundy BN, Long SA, Bluestone JA, DiMeglio LA, Dufort MJ, Gitelman SE, Gottlieb PA, Krischer JP, Linsley PS, Marks JB, Moore W, Moran A, Rodriguez H, Russell WE, Schatz D, Skyler JS, Tsalikian E, Wherrett DK, Ziegler AG, Greenbaum CJ; Type 1 Diabetes TrialNet Study Group. An Anti-CD3 Antibody, Teplizumab, in Relatives at Risk for Type 1 Diabetes. N Engl J Med. 2019 Aug 15;381(7):603-613. doi: 10.1056/NEJMoa1902226. Epub 2019 Jun 9. PMID 31180194
- [Background] Hummel S, Carl J, Friedl N, Winkler C, Kick K, Stock J, Reinmuller F, Ramminger C, Schmidt J, Lwowsky D, Braig S, Dunstheimer D, Ermer U, Gerstl EM, Weber L, Nellen-Hellmuth N, Bramswig S, Sindichakis M, Tretter S, Lorrmann A, Bonifacio E, Ziegler AG, Achenbach P; Fr1da Study Group. Children diagnosed with presymptomatic type 1 diabetes through public health screening have milder diabetes at clinical manifestation. Diabetologia. 2023 Sep;66(9):1633-1642. doi: 10.1007/s00125-023-05953-0. Epub 2023 Jun 17. PMID 37329450
- [Background] Barker JM, Goehrig SH, Barriga K, Hoffman M, Slover R, Eisenbarth GS, Norris JM, Klingensmith GJ, Rewers M; DAISY study. Clinical characteristics of children diagnosed with type 1 diabetes through intensive screening and follow-up. Diabetes Care. 2004 Jun;27(6):1399-404. doi: 10.2337/diacare.27.6.1399. PMID 15161795
- [Background] Krischer JP, Liu X, Vehik K, Akolkar B, Hagopian WA, Rewers MJ, She JX, Toppari J, Ziegler AG, Lernmark A; TEDDY Study Group. Predicting Islet Cell Autoimmunity and Type 1 Diabetes: An 8-Year TEDDY Study Progress Report. Diabetes Care. 2019 Jun;42(6):1051-1060. doi: 10.2337/dc18-2282. Epub 2019 Apr 9. PMID 30967432
- [Background] McQueen RB, Geno Rasmussen C, Waugh K, Frohnert BI, Steck AK, Yu L, Baxter J, Rewers M. Cost and Cost-effectiveness of Large-scale Screening for Type 1 Diabetes in Colorado. Diabetes Care. 2020 Jul;43(7):1496-1503. doi: 10.2337/dc19-2003. Epub 2020 Apr 23. PMID 32327420
- [Background] American Diabetes Association Professional Practice Committee. 2. Diagnosis and Classification of Diabetes: Standards of Care in Diabetes-2024. Diabetes Care. 2024 Jan 1;47(Suppl 1):S20-S42. doi: 10.2337/dc24-S002. PMID 38078589
- [Background] Krischer JP, Lynch KF, Schatz DA, Ilonen J, Lernmark A, Hagopian WA, Rewers MJ, She JX, Simell OG, Toppari J, Ziegler AG, Akolkar B, Bonifacio E; TEDDY Study Group. The 6 year incidence of diabetes-associated autoantibodies in genetically at-risk children: the TEDDY study. Diabetologia. 2015 May;58(5):980-7. doi: 10.1007/s00125-015-3514-y. Epub 2015 Feb 10. PMID 25660258
- [Background] Ziegler AG, Rewers M, Simell O, Simell T, Lempainen J, Steck A, Winkler C, Ilonen J, Veijola R, Knip M, Bonifacio E, Eisenbarth GS. Seroconversion to multiple islet autoantibodies and risk of progression to diabetes in children. JAMA. 2013 Jun 19;309(23):2473-9. doi: 10.1001/jama.2013.6285. PMID 23780460
- [Background] Insel RA, Dunne JL, Atkinson MA, Chiang JL, Dabelea D, Gottlieb PA, Greenbaum CJ, Herold KC, Krischer JP, Lernmark A, Ratner RE, Rewers MJ, Schatz DA, Skyler JS, Sosenko JM, Ziegler AG. Staging presymptomatic type 1 diabetes: a scientific statement of JDRF, the Endocrine Society, and the American Diabetes Association. Diabetes Care. 2015 Oct;38(10):1964-74. doi: 10.2337/dc15-1419. PMID 26404926
- [Background] TEDDY Study Group. The Environmental Determinants of Diabetes in the Young (TEDDY) Study. Ann N Y Acad Sci. 2008 Dec;1150:1-13. doi: 10.1196/annals.1447.062. PMID 19120261
- [Background] Besser REJ, Bell KJ, Couper JJ, Ziegler AG, Wherrett DK, Knip M, Speake C, Casteels K, Driscoll KA, Jacobsen L, Craig ME, Haller MJ. ISPAD Clinical Practice Consensus Guidelines 2022: Stages of type 1 diabetes in children and adolescents. Pediatr Diabetes. 2022 Dec;23(8):1175-1187. doi: 10.1111/pedi.13410. Epub 2022 Sep 30. No abstract available. PMID 36177823
- [Background] Besser REJ, Ng SM, Gregory JW, Dayan CM, Randell T, Barrett T. General population screening for childhood type 1 diabetes: is it time for a UK strategy? Arch Dis Child. 2022 Sep;107(9):790-795. doi: 10.1136/archdischild-2021-321864. Epub 2021 Nov 5. PMID 34740879
- See also: Published protocol — https://wellcomeopenresearch.org/articles/9-601